CLINICAL TRIAL: NCT04067466
Title: Effect on Appetite Satisfaction and Short-term Satiety of Different Plant Compositions in the Adolescent Age Group
Brief Title: Appetite Satisfaction and Short-term Satiety of Different Plant Compositions in the Adolescent Age Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorios Ordesa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: VEGYDOWN-15 (B)
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Satiety; Appetite
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber product (Experimental): Fiber product: Inulin, maltodextrin, gum guar, plum powder
  Interventions: Dietary Supplement: Fiber product
- Control product (Placebo Comparator): Maltodextrin, plum powder
  Interventions: Dietary Supplement: Control product

INTERVENTIONS:
Dietary Supplement: Fiber product — Fiber product with inulin, maltodextrin, gum guar and plum powder.
  Arms: Fiber product
Dietary Supplement: Control product — Placebo product with maltodextrin and plum powder
  Arms: Control product

SUMMARY:
This study evaluates the satiating effect of two types of food supplements made from various types of fibres in the subsequent intake of other foods, in satiety, and in the regulation of hormones

DETAILED DESCRIPTION:
This study assessing the effect on appetite satisfaction and short-term satiety of different plant compositions in the adolescent age segment wants to assess the satiating effect of two types of food supplements made with various types of fibers (inulin, maltodextrins, guar gum and dehydrated plums) in the subsequent intake of other foods, in satiety, and in the regulation of hormones (ghrelin, leptin and insulin) and other peptides involved in the mechanisms of satiety

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 15 and 30 years old.
* Subjects with IMC<25 kg/m2
* Subjects who have a habit of having breakfast, lunch and dinner every day
* Subjects who are willing to comply with the study procedures

Exclusion Criteria:

* Subjects taht are taking any medicines that affect the appetite or food intake
* Presence of endocrine-metabolic diseases
* Eating disorders
* Subjects who are following a special diet
* Subjects who have changed their body weight by more than 10% in the last three months prior to the study
* Subjects who follow a restrictive dietary pattern such as vegetarians, gluten-free diets, weight loss diets, etc.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of satiety using objective methods (blood analysis) | Change from week 1 to week 2
  Biochemistry : glucose, urea, BUN, creatinin (all in mg/dL)
Assessment of satiety (blood analysis) | Change from week 1 to week 2
  Biochemistry : GOT and GPT (UI/L)
Assessment of satiety using a subjective method (visual analogue scale) | Change from week 1 to week 2
  The perceived feeling of satiety will be measured using the 100mm "Visual Analogue Scale" labeled at a far end with a "mark" to the left of "extremely hungry", and on the other with an "extremely satiated"."

CONTACTS AND LOCATIONS:
Overall Officials: Luis Moreno Aznar, Principal Investigator — Universidad de Zaragoza
Locations (1):
- GENUD Research Group, Universidad de Zaragoza, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No